CLINICAL TRIAL: NCT03245567
Title: Implementation and Evaluation of a Perceptual Learning Module on the Visual Estimation of Left Ventricular Ejection Fraction Using Transesophageal Echocardiography
Brief Title: Implementation and Evaluation of a Perceptual Learning Module on Visual Estimation of LVEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17.119
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Medical Education
MeSH Terms: interventions — Lead

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre, post, delayed test (Experimental): Participants will not do the PLM, but will perform a pretest, a posttest and a delayed test at 6 months
  Interventions: Other: Pre, post, delayed test
- PLM group (pre, post, delayed test, PLM) (Experimental): Participants will do a pretest, the PLM, a posttest and a delayed test at 6 months
  Interventions: Other: PLM; Other: Pre, post, delayed test

INTERVENTIONS:
Other: PLM — Participants will take the PLM on the visual estimation of LVEF. They will also take a pretest, a post-test and a delayed test at 6 months.
  Arms: PLM group (pre, post, delayed test, PLM)
Other: Pre, post, delayed test — Participants will perform a pretest, a posttest and a delayed test at 6 months.

SUMMARY:
This study is designed to:

1. Implement a Web platform intended to host perceptual learning modules (PLMs)
2. Implement and assess a PLM designed to improve the capacity of first-year residents and fourth-year medical students to visually estimate the left ventricular ejection fraction (LVEF) with transesophageal echocardiography (TEE) images.

The hypothesis of the study is that the PLM will improve the visual assessment of LVEF by TEE in junior residents and medical students.

DETAILED DESCRIPTION:
TEE is increasingly used for perioperative diagnosis and monitoring. However, learning TEE may be long and difficult: guidelines suggest that learners perform and interpret hundreds of TEE exams during their training. Even if this learning process has been used successfully for many years, it has important limitations, especially in the context of an ever-increasing number of trainees: access to patients and TEE experts is limited, and the extensive period of time required to train is also a problem.

Simulators have gained popularity as tools for teaching echocardiography, showing benefits mostly regarding probe handling and image acquisition. Some simulators may also be useful to replicate some diseases, but most simulators can only replicate a limited variety of diseases, and mostly typical presentations. This is an important limitation when it comes to teaching image interpretation. In order to develop their expertise, trainees have to be exposed to a wide range of normal variations and to more subtle abnormalities.

PLMs represent an alternative modality to teach image interpretation, and are already used in other fields. PLMs are online tools created to enhance the development of pattern recognition, a skill required to efficiently interpret TEE images. With PLMs, learners observe a series of images or videoclips and must answer a question about each image in a short period of time. Each answer is followed by an immediate feedback (the correct answer). By observing a large number of images online and by receiving systematic and expert feedback, the trainee quickly learns to extract efficiently the required information from the image.

This study will aim to evaluate the effects of a PLM on the ability of junior residents and medical students to correctly estimate visually the left ventricular ejection faction using TEE images.

Methods:

A team of experienced programmers will develop a Web platform, which will allow the identification of both participants and TEE experts, manage the consent process, host the tests used to assess the participants' expertise and the PLM itself, as well as manage the TEE images and the study data.

The pilot study designed to assess the impact of the PLM on the visual estimation of LVEF will be composed of the following steps:

1. selection and validation of TEE cases,
2. development of two versions of a test and of the PLM,
3. analysis of the impact of the PLM on participants' performance vs a control group.

Each TEE case used in this study will comprise 3 short video loops containing the following standardised echocardiographic views:

* midesophageal four chamber view
* midesophageal two chamber view
* midesophageal long axis view

Prior to inclusion in the study, each case will be anonymized and then validated by two cardiologists expert in TEE interpretation. Only cases where the visual estimation of the LVEF provided independently by the two TEE experts will differ by no more than 10% will be used. Two different sets of validated images will then be created.

The first set will be comprised of two groups of 20 validated cases (total of 40 cases). These cases will be used to create two versions of a test used to assess participants' expertise in the visual estimation of LVEF at different stages in the research protocol. These cases will not be part of the PLM.

The second set will be comprised of 96 validated cases destined to the PLM. The PLM is designed not to assess the participants' expertise, but to develop their ability to estimate LVEF.

When taking a test on the platform, participants will see the three short video loops of each case simultaneously on the screen for a maximum of 20 seconds, and will then have to provide an estimation of the LVEF. Each answer will be followed immediately by another case, and no feedback will be provided.

When doing the PLM, participants will see the three short video loops of each case simultaneously on the screen for a maximum of 20 seconds, and will then have to provide an estimation of the LVEF. However, each answer will be followed by feedback in the form of the average value of the experts' visual estimates of LVEF. This sequence of "case visualisation - participant estimation - expert feedback" will be repeated 96 times during this PLM.

Residents and medical students will be randomised by the platform to a Control Group and a PLM group. Both groups will participate in two on-line sessions. During the first session, demographic and clinical experience data will be collected. All participants will also perform a pretest to measure their baseline ability to estimate LVEF. Then only the participants randomised to the PLM group will do the PLM. All participants will do a posttest at the end of the first session. Six months later, all participants will return for a second session to perform the delayed test.

At the end of the study, participants of the Control group will be allowed to complete the PLM if they wish to.

ELIGIBILITY:
Inclusion Criteria:

* Residents in their first year of training or fourth-year medical students having access to a computer with a high speed internet connection
* Residents or medical students with no significant experience in echocardiography

Exclusion Criteria:

* Smartphones and tablets will not be acceptable to perform the tests due to their smaller screens
* Residents or medical students having significant experience with transthoracic or transesophageal echocardiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in accuracy of LVEF estimation in the Control group versus the PLM group | At baseline (pretest) and on the immediate posttest
  For each case, the absolute difference between the participant and the experts' estimation of LVEF is calculated. Participant's accuracy is defined as the average of absolute differences for all cases in the test

SECONDARY OUTCOMES:
Change in accuracy of LVEF estimation in the Control group versus the PLM group | At baseline (pretest) and on the delayed post-test (6 months)
  For each case, the absolute difference between the participant and the experts' estimation of LVEF is calculated. Participant's accuracy is defined as the average of absolute differences for all cases in the test
Change in the mean response time in seconds to the different tests in the Control group versus the PLM group | At baseline (pretest), on an immediate posttest, and on the delayed test at 6 months
The evolution of the participants' accuracy in LVEF estimation during the PLM | During the PLM, at the end of the first on-line session
  For each case, the absolute difference between the participant and the experts' estimation of LVEF is calculated. The 96 cases in the PLM will be placed in 8 groups of 12 cases. Participant's accuracy for a group is defined as the average of absolute differences for all cases in that group.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Robitaille, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Champagne P, Girard F, Cyr V, Romanelli G, Ruel M, Todorov A, Robitaille A. The impact of a perceptual learning module on novices' ability to visually estimate left ventricular ejection fraction by transesophageal echocardiography: a randomized controlled study. Can J Anaesth. 2021 Oct;68(10):1527-1535. doi: 10.1007/s12630-021-02066-3. Epub 2021 Jul 28. PMID 34319575